CLINICAL TRIAL: NCT05400876
Title: Phase Ib Clinical Trial to Evaluate the Efficacy and Safety of TQB2618 Injection Combined With Penpulimab in Patients With Relapsed or Refractory Lymphoma
Brief Title: To Evaluate the Safety and Efficacy of TQB2618 Injection Combined With Penpulimab in the Treatment of Patients With Relapsed and Refractory Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-AK105-Ib-01
Record Dates: First submitted 2022-05-16; First posted 2022-06-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-06

CONDITIONS: Relapsed/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2618 injction+penpulimab injection (Experimental): TQB2618 injection with penpulimab injection, 21 days as a treatment cycle
  Interventions: Drug: TQB2618 injection; Drug: Penpulimab injection

INTERVENTIONS:
Drug: TQB2618 injection — TQB2618 injection is an inhibitor of T cell immunoglobulin and mucin domain-containing protein 3 (TIM3)
Drug: Penpulimab injection — Penpulimab is an inhibitor of programmed cell death protein 1 (PD-1)

SUMMARY:
This is a two-phase, open-label Phase Ib clinical trial to evaluate the safety and efficacy of TQB2618 injection combined with Penpulimab in patients with relapsed and refractory lymphoma

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects with pathologically proven with relapsed or refractory lymphoma and with disease progression during or after the last treatment or no objective response confirmed after adequate treatment.
* 2 Cohort 1: Subjects with Classical Hodgkin lymphoma (cHL) who had previously received at least twice systemic therapy and are resistant to PD-1 or PD-L1.
* 3 Cohort 2: Subjects with B lymphocyte non-Hodgkin lymphoma (B-NHL) who had previously received at least twice systemic therapy containing anti-CD20-targeted therapy.
* 4 Cohort 3：Subjects with T lymphocyte non-Hodgkin lymphoma (T-NHL) who had previously received at least one systemic therapy.
* 5 Subjects with measurable lesions as defined by Lugano2014.
* 6 Aged 18-75 years ; Eastern Cooperative Oncology Group (ECOG) score:0 ~ 1; Expected survival ≥3 months.
* 7 Laboratory indicators meet the requirements.
* 8 Subjects voluntarily joined the study and signed the informed consent form.
* 9 Non-pregnant or non-breastfeeding women; Negative pregnancy subjects.

Exclusion Criteria:

* 1 Subjects who have developed or is currently suffering from other malignancies within 3 years, with the exception of cured skin basal cell carcinoma and cervical carcinoma in situ.
* 2 Subjects who have not recovered to ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 due to the adverse event of prior therapy.
* 3 Subjects with significant surgery or significant traumatic injury within 28 days before first injection (excluding needle biopsy or endoscopic biopsy).
* 4 Subjects with long-term unhealed wounds or fractures.
* 5 Subjects with the high risk of bleeding or bleeding history or subjects with bleeding event (≥Common Terminology Criteria for Adverse Events Grade 3) within 4 weeks before first injection.
* 6 Subjects with arterial/venous thrombosis within 6 months.
* 7 Subjects with a history of psychotropic substance abuse who cannot be withdrawn or have mental disorders.
* 8 Subjects with any severe and/or uncontrolled disease.
* 9 subjects with lymphoma originating from Central Nervous System, high-grade B-cell lymphoma or hemophagocytic syndrome during screening period.
* 10 Subjects with violating Central Nervous System (CNS) .
* 11 Subjects with allogeneic hematopoietic stem cell transplantation.
* 12 Subjects with autologous hematopoietic stem cell transplantation or Chimeric Antigen Receptor T-Cell Immunotherapy(CAR-T) within 3 months before first injection.
* 13 Subjects with other factors that might cause the study to be terminated halfway per the judgement of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
dose limiting toxicity/DLT | From the first injection up to 3 weeks
  The relevant adverse reactions occurred within the first cycle
recommended phase II dose/RP2D | From the first injection up to 6 weeks
  The dose of TQB2618 injection which is recommended to use during phase II clinical trial
Overall response rate (ORR) based on 2014 Lugano | From the first injection up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
complete remission rate/CRR | From the first injection up to 96 weeks
  Percentage of participants achieving complete response
Disease control rate/DCR | From the first injection up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | From the first injection up to 120 weeks
  The time when the participants first achieved CR or PR to disease progression or death from any cause.
Progression-free survival (PFS) | Up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
  cause.
  cause. PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival/OS | From date of randomization until the death from any cause, assessed up to 120 weeks
  OS defined as the time from randomization until the death from any cause
Peak time/Tmax | Cycle 1 day 1 Before administration, 30 minuets,4,8,24,48,144,312 hours after minuets, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1, Cycle 5 day 1, Cycle 6 day 1, Cycle 7 day 1, Cycle 8 day 1 before and 30 minutes after administration.each cycle 21 days
  The time to peak concentration
Peak concentration (Cmax) | Cycle 1 day 1 Before administration, 30 minuets,4,8,24,48,144,312 hours after minuets, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1, Cycle 5 day 1, Cycle 6 day 1, Cycle 7 day 1, Cycle 8 day 1 before and 30 minutes after administration.（each cycle 21 days）
  Maximum plasma drug concentration
Half-life /T1/2 | Cycle 1 day 1 Before administration, 30 minuets,4,8,24,48,144,312 hours after minuets, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1, Cycle 5 day 1, Cycle 6 day 1, Cycle 7 day 1, Cycle 8 day 1 before and 30 minutes after administration.（each cycle 21 days)
  The time it takes for the drug's concentration in the body to drop by half
Receptor Occupancy/RO | Cycle 1 day 1, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1, Cycle 5 day 1, Cycle 6 day 1, Cycle 7 day 1, Cycle 8 day 1 before administration and 30 minutes after administration and the day of disease progression（each cycle 21 days)
  The extent to which antibody drugs occupy cell surface targets
Incidence of Anti-Drug antibody and neutralizing antibodies | Cycle 1 day 1, Cycle 2 day 1, Cycle 4 day 1, Cycle 8 day 1,before administration and 30, 90 days after the last administration（each cycle 21 days)
  The incidence of anti-drug antibody and neutralizing antibodies after administration of TQB2618 and penpulimab
Adverse event rate | Baseline up to 96 weeks
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China